CLINICAL TRIAL: NCT06247748
Title: Evaluation of the Effects of Exendin-4 Fc Fusion Protein (JY09) Injection on the Pharmacokinetic Profiles of Metformin Hydrochloride Tablets, Rosuvastatin Calcium Tablets, and Digoxin Tablets and on the QT Interval in Overweight Chinese Subjects
Brief Title: Influence of JY09 on Pharmacokinetics of Metformin , Rosuvastatin , and Digoxin and the QT Interval Study in Overweight Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing Dongfang Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: dfbt-jy09-ow-2023-101
Record Dates: First submitted 2024-01-22; First posted 2024-02-08 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2; Overweight
Keywords: JY09; QT Interval
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight | interventions — Injections; Metformin; Rosuvastatin Calcium; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exendin-4 Fc fusion protein (JY09) injection (Experimental): D22 received a single subcutaneous abdominal injection of 1.2 mg of JY09 injection after completion of PK blood sampling; D29 to D78 received continuous subcutaneous abdominal injections of 2.4 mg of JY09 injection in the morning, once weekly (total of 8 administrations). All doses were to be administered within 3 min.
  Interventions: Drug: Exendin-4 Fc fusion protein (JY09) injection; Drug: Metformin Hydrochloride tablet; Drug: Rosuvastatin calcium tablets; Drug: Digoxin tablet

INTERVENTIONS:
Drug: Exendin-4 Fc fusion protein (JY09) injection — D22 received a single subcutaneous abdominal injection of 1.2 mg of JY09 injection after completion of PK blood sampling; D29, D36, D43, D50, D57, D64, D71, and D78 subjects returned to the study center to receive a subcutaneous abdominal injection of 2.4 mg of JY09 injection(total of 8 administrations).All doses were to be administered within 3 min.
  Other Names: JY09
Drug: Metformin Hydrochloride tablet — D1 to D4 continuous oral administration of 0.5 g metformin hydrochloride tablets twice daily (D4 was administered only in the morning, with a total of 7 administrations) for a washout period of 96 h;0.5 g metformin hydrochloride tablets orally twice a day continuously from D85 to D88 (D88 was given only in the morning, for a total of 7 doses).
  Other Names: Metformin
Drug: Rosuvastatin calcium tablets — D8 received a single oral administration of 10 mg of Rosuvastatin calcium tablets in the morning, with a washout period of 168 h,and 10 mg Rosuvastatin calcium tablets orally at 72 h ± 0.5 h (D95) after JY09 administration.
  Other Names: Rosuvastatin
Drug: Digoxin tablet — D15 received a single oral administration of 0.25 mg digoxin tablets in the morning, with a washout period of 168 h,oral 0.25 mg digoxin tablets 72 h±0.5 h after JY09 administration (D102)
  Other Names: digoxin

SUMMARY:
This trial is conducted in china. The aim of the trial is as follows:

* To assess the effect of multiple subcutaneous injections of JY09 injection on the pharmacokinetic (PK) profile of multiple oral doses of metformin hydrochloride tablets, a single oral dose of Rosuvastatin calcium tablets, or digoxin tablets in overweight Chinese subjects;
* To assess the effect of multiple subcutaneous injections of JY09 injection on QT interval in overweight Chinese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age: Overweight subjects with full capacity for civil behavior who are ≥ 18 years old and ≤ 45 years old (the ratio of the number of subjects of either sex is not less than 1/3).
2. Body weight: men ≥ 50.0 kg, women ≥ 45.0 kg, body mass index (BMI) ≥ 24.0 kg/m2 and ≤ 28.0 kg/m2 , BMI = weight (kg)/height (m2 ).
3. Those who do not plan to have children in the last 6 months, do not plan to donate sperm/eggs, and are willing to use effective contraception for 6 months after the end of dosing.
4. Fully understand the trial and possible adverse effects, have the ability to communicate normally with the investigator, as well as comply with study requirements, follow protocol procedures and limitations, and be able to visit on time.
5. Understand the content of the informed consent form, agree to participate in this trial and voluntarily sign the consent form.

Exclusion Criteria:

1. A clear history of central nervous system, cardiovascular system, renal, hepatic, pulmonary, metabolic, and musculoskeletal disorders or other notable diseases.
2. Individuals with gastrointestinal disorders, such as history of hepatobiliary disease, history of gastrointestinal disease, history of gastrointestinal surgery (except appendectomy) or history of chronic pancreatitis or idiopathic acute pancreatitis, and those with habitual diarrhea.
3. Previous tip-twisting ventricular tachycardia or other risk factors that can lead to malignant arrhythmias, or a family history of first-degree relatives (i.e., biological parents, siblings, or children) with short QT syndrome, long QT syndrome, unexplained sudden death, drowning, or sudden infant death syndrome in young adulthood (less than/equal to 40 years of age), or cardiac conduction block.
4. Have disorders of electrolyte metabolism such as hyperkalemia, hypokalemia, hypomagnesemia, hypomagnesemia, hypercalcemia or hypocalcemia.
5. If the results of vital signs (blood pressure, pulse, respiration, temperature) are abnormal and clinically significant, a retest is allowed to confirm the results if they are abnormal, and the abnormal values of each vital sign.
6. Physical examination, laboratory tests, 12-lead electrocardiogram (ECG), abdominal ultrasound, calcitonin and chest radiographs (orthopantomograms) suggesting the presence of abnormalities judged by the investigator to be clinically significant (retesting was allowed once).
7. Smokers who smoked an average of more than 5 cigarettes per day in the 3 months prior to screening or who could not give up smoking during their participation in the trial or who had a positive smoke test.
8. Those who have participated in other clinical trials as a subject within 3 months prior to screening.
9. Those who donated blood or blood products ≥400 mL within 3 months prior to screening.
10. Those who cannot tolerate venipuncture and have a history of needle and blood sickness.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
The Metformin Peak Concentration (Cmax ) | During a dosing interval (0-36 hours) after the last of 7 repeated doses of metformin without JY09 exposure (Day 4) and at JY09 steady state (Day 88)
  The peak concentration(Cmax） is the highest level of plasma concentration that occurs after administration.This parameter is an important index to reflect the absorption rate and degree of drug in vivo.
Area under the Metformin blood concentration-time curve | During a dosing interval (0-36 hours) after the last of 7 repeated doses of metformin without JY09 exposure (Day 4) and at JY09 steady state (Day 88)
  AUC refers to the area under the drug time curve, which is the area surrounded by the pharmacokinetic blood concentration curve to the time axis. This parameter is an important index to evaluate the degree of drug absorption, reflecting the exposure characteristics of drugs in vivo.
The Rosuvastatin Peak Concentration (Cmax ) | From time 0 to 96 hours after a single dose of Rosuvastatin without JY09 exposure (Day 8) and at JY09 steady state (Day 95)
  The peak concentration(Cmax） is the highest level of plasma concentration that occurs after administration.This parameter is an important index to reflect the absorption rate and degree of drug in vivo.
Area under the Rosuvastatin blood concentration-time curve | From time 0 to 96 hours after a single dose of Rosuvastatin without JY09 exposure (Day 8) and at JY09 steady state (Day 95)
  Area under curve(AUC) refers to the area under the drug time curve, which is the area surrounded by the pharmacokinetic blood concentration curve to the time axis. This parameter is an important index to evaluate the degree of drug absorption, reflecting the exposure characteristics of drugs in vivo.
The Digoxin Peak Concentration (Cmax ) | From time 0 to 168 hours after a single dose of Digoxin without JY09 exposure (Day 15) and at JY09 steady state (Day 102)
  The peak concentration(Cmax） is the highest level of plasma concentration that occurs after administration.This parameter is an important index to reflect the absorption rate and degree of drug in vivo.
Baseline-corrected difference of Corrected QT interval after multiple subcutaneous injections of JY09 injection | From time 0 to 72 hours after a single dose of JY09 (Day 22) and at JY09 steady state (Day 92)
  Corrected QT interval is a QT interval adjusted by heart rate, which is an index of cardiac depolarization and repolarization

SECONDARY OUTCOMES:
Safety endpoint-Adverse events | From baseline (Day -1) to follow-up (Day 123)
  All adverse medical events occurring after the subject receives the experimental drug, which may be manifested as symptoms, signs, diseases, or abnormalities in laboratory tests, but may not necessarily have a causal relationship with the experimental drug.
Vital signs-Blood pressure | From baseline (Day -1) to follow-up (Day 123)
  Blood pressure includes systolic and diastolic blood pressure.
Vital signs-Pulse | From baseline (Day -1) to follow-up (Day 123)
  Pulse refers to the pulsation formed in the arteries when the heart contracts, due to the flow of blood from the heart into the arteries. Pulse is one of the vital signs of human body, and it is an important index to measure heart rate and blood pressure.
Vital signs-Respiration | From baseline (Day -1) to follow-up (Day 123)
  Respiration refers to the process of gas exchange between the body and the outside world.
Physical examination | From baseline (Day -1) to follow-up (Day 123)
  Include general condition, skin, neck (including thyroid), head (including eyes, ears, nose, throat), chest, abdomen, back, lymph nodes, limbs, and nervous system.
Laboratory tests-Routine blood | From baseline (Day -1) to follow-up (Day 123)
  Blood routine refers to the examination of blood conditions and diseases by observing the changes in the number and morphological distribution of blood cells.
Laboratory tests-Blood biochemistry | From baseline (Day -1) to follow-up (Day 123)
  Blood biochemical examination can determine the content of sugars, lipids, hormones, ions and other substances in the blood, and provide help for the diagnosis and treatment of diseases.
Laboratory tests-Urine routine | From baseline (Day -1) to follow-up (Day 123)
  Urine routine is of great significance not only for the observation of the curative effect of the diagnosis of urinary system diseases, but also for the diagnosis and prognosis of other system diseases.
Laboratory tests-coagulation function | From baseline (Day -1) to follow-up (Day 123)
  The coagulation function test is mainly to find out whether the clotting factors in the patient's body are abnormal.
12-lead electrocardiogram (ECG) | From baseline (Day -1) to follow-up (Day 123)
  Electrocardiogram (ECG) is an objective index of the occurrence, propagation and recovery of cardiac excitation. It is used for the examination of various arrhythmias, ventricular and atrial hypertrophy, myocardial infarction, arrhythmia, myocardial ischemia and other diseases.
Immunogenicity | From baseline (Day -1) to follow-up (Day 123)
  Immunogenicity refers to the performance that can cause an immune response, that is, the antigen can stimulate specific immune cells, so that immune cells activation, proliferation, differentiation, and eventually produce immune effecting substances antibodies and sensitized lymphocytes.

OTHER OUTCOMES:
Area Under the Effect Curve from time 0 to the last measurable concentration (AUEC0-t ) | From time 0 to 240 minutes after Oral glucose(Day21) and Oral glucose(Day84).
  AUEC0-t is a Pharmacodynamics -related endpoint for glucose, C-peptide and insulin in the Oral glucose tolerance test (OGTT),which reflects the amount of exposure to the effect.
The Peak Effect Concentration(ECmax） | From time 0 to 240 minutes after Oral glucose(Day21) and Oral glucose(Day84).
  ECmax is a Pharmacodynamics -related endpoint for glucose, C-peptide and insulin in the Oral glucose tolerance test (OGTT),which reflects the maximum effective concentration.
Maximum Effect Time(ETmax ) | From time 0 to 240 minutes after Oral glucose(Day21) and Oral glucose(Day84).
  ETmax is a Pharmacodynamics -related endpoint for glucose, C-peptide and insulin in the Oral glucose tolerance test (OGTT),which reflects the time of the first maximum effect.
(AUEC0-t after JY09 administration - AUEC0-t before JY09 administration)/AUEClast before JY09 administration ×100%(Δ%AUEC0-t) | From time 0 to 240 minutes after Oral glucose(Day21) and Oral glucose(Day84).
  Δ%AUEC0-t is a Pharmacodynamics -related endpoint for glucose, C-peptide and insulin in the Oral glucose tolerance test (OGTT), which reflects changes in the amount of effect exposure before and after administration.
(post-administration Maximum Effect(Emax)- pre-administration Maximum Effect(Emax))/pre-administration Maximum Effect(Emax)×100%(Δ%Emax ) | From time 0 to 240 minutes after Oral glucose(Day21) and Oral glucose(Day84).
  Δ%Emax is a Pharmacodynamics -related endpoint for glucose, C-peptide and insulin in the Oral glucose tolerance test (OGTT), which reflects changes in maximum effects before and after administration.
Body fat mass | Day19 or Day20,Day103 or Day104.
  Body fat mass refers to the amount of fat in a person's body.
Body fat percentage | Day19 or Day20,Day103 or Day104.
  Body fat percentage refers to fat content as a percentage of total body weight.
Fat-free weight | Day19 or Day20,Day103 or Day104.
  Fat-free weight refers to the body weight after the removal of fat, also known as lean body weight, is the weight of other body components other than fat.
Skeletal muscle mass | Day19 or Day20,Day103 or Day104.
  Skeletal muscle mass is the percentage of skeletal muscle in the body, and can be used to determine health status.
Waist-to-hip ratio | Day19 or Day20,Day103 or Day104.
  Waist-to-hip ratio is the ratio between waist and hip circumference and is an important indicator of central obesity.
Visceral fat area | Day19 or Day20,Day103 or Day104.
  Visceral fat area is an indicator used to assess the degree of abdominal obesity in an individual, and it can be measured in a number of ways, such as CT (computed tomography) or MRI (magnetic resonance imaging). This area of adipose tissue around the abdomen is associated with the risk of a number of chronic diseases such as heart disease and diabetes.
Pharmacodynamically relevant plasma endogenous markers（If necessary） | From time 0 to 72 hours after a single dose of JY09 (Day 22) and at JY09 steady state (Day 92) and Day21，Day29，Day43，Day83
  The investigator will use JY09 PK residual or backup plasma samples from this trial to assay efficacy-related endogenous marker concentrations to support individualized dosing of JY09.
Pharmacodynamically relevant plasma metabolomics(if necessary) | From time 0 to 72 hours after a single dose of JY09 (Day 22) and at JY09 steady state (Day 92) and Day21，Day29，Day43，Day83
  The investigator will use JY09 PK residual or backup plasma samples from this trial to assay efficacy-related metabolomics to support individualized dosing of JY09.
Blood Cell Genotype Characterization (if necessary) | Day21，Day29，Day43，Day83
  Blood cell samples after centrifugation at each time point of the immunogenicity assay were retained for each subject so that they could be used for genotypic testing at a later stage, if necessary, to support individualized dosing of JY09.
Bacteria genus | Day21 or Day22,Day84 or Day85
  Species of bacteria in intestinal flora.
Relative abundance | Day21 or Day22,Day84 or Day85
  Relative abundance of genera and strains of bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital drug clinical trial Institute, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No